CLINICAL TRIAL: NCT01837316
Title: A Randomized, Double-blind, Placebo-controlled Cross-over Study to Determine the Bronchodilator Effect of a Single Dose of Fluticasone Furoate (FF)/ Vilanterol (VI) 100/25 mcg Combination Administered in the Morning in Adult Patients With Asthma
Brief Title: A Study to Assess the Bronchodilator Effect of a Single Dose of Fluticasone Furoate (FF)/ Vilanterol (VI) 100/25 Micrograms (mcg) Combination When Administered in Adult Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116592
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: pharmacodynamics; FF/VI; asthma; duration of action
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/VI (Experimental): A single dose inhalation of FF/VI 100/25 mcg in the morning
  Interventions: Drug: FF/VI 100/25 mcg
- Placebo (Placebo Comparator): A single dose inhalation of matching placebo in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FF/VI 100/25 mcg — First strip: Fluticasone furoate inhalation powder blended with lactose, 100 mcg per blister
  Arms: FF/VI
Drug: Placebo — First strip: Inhalation powder of lactose
  Arms: Placebo

SUMMARY:
The study will be a randomized, double-blind, placebo controlled cross-over study in 32 adult subjects with moderately severe asthma. In this study the bronchodilator effect of a single morning dosing of FF/VI combination 100/25 mcg will be determined by spirometry. After the screening the subject will be randomized and will be assigned to one of two treatment sequences (AB or BA, where A is placebo and B is FF/VI 100/25 mcg). Between the two treatment periods there will be a washout period of 7-14 days. A serial forced expiratory volume in one second (FEV1) measurements will be taken at 15, 30 minutes, 1, 2, 4, 12, 24, 36, 48, 60 and 72 hours post dose. Safety assessments will include vital signs, electrocardiograms (ECGs), adverse event (AE) monitoring and laboratory safety tests however, these will not constitute study endpoints. The results of the study will provide supporting information to prescribers on the bronchodilator effect of FF/VI over 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Asthma: A doctor diagnosis of asthma.
* Age of subject: 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Severity of Disease: A screening pre-bronchodilator FEV1 >=60% of predicted.
* Reversibility of Disease: Demonstrated presence of reversible airway disease at screening.
* Current Therapy: On inhaled corticosteroid (ICS) with or without a SABA for at least 12 weeks prior to screening. Able to stop current Short-Acting Beta2-Agonists (SABA) and replace with albuterol/salbutamol inhaler
* Body weight and BMI: Body weight >=50 kilogram (kg) and Body Mass Index (BMI) within the range 19.0 to 29.9 kilogram per square meter (kg/m^2) (inclusive).
* Gender: Male or female. A female subject is eligible to participate if she is of:

Non-childbearing potential. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

Child-bearing potential and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.

* Liver criteria: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2x Upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Consent: Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A history of life-threatening asthma.
* Other significant pulmonary diseases: pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening that; led to a change in asthma management OR in the opinion of the Investigator, is expected to affect the subject's asthma status OR the subject's ability to participate in the study.
* Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of screening or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to screening.
* Concomitant Medications: Use of the medications, ICS were prohibited for each study period from 24 hours prior to dosing to 72 hours after dosing; Long acting beta agonist (LABA), leukotriene receptor antagonist (LTRA) or long acting muscarinic anatagonist (LAMA) were prohibited for 12 weeks prior to screening; High doses of an ICS were prohibited for 8 weeks prior to screening; Oral steroids were prohibited for 12 weeks prior to screening; Potent CYPP3A4 inhibitors were prohibited within 4 weeks prior to dosing. The following medications may not be used during the study from first dosing to the end of period 2 inclusive: Anticonvulsants, Polycyclic antidepressants, β-adrenergic blocking agents, Phenothiazines and Monoamine oxidase (MAO) inhibitors.
* Other concurrent Diseases/Abnormalities: A subject has any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the study results if the condition/disease exacerbated during the study.
* Oropharyngeal examination: A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis at screening.
* Pregnancy and Lactating Females:Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at screening or by positive urine hCG test prior to dosing. Lactating females.
* Allergies: Milk Protein Allergy: History of severe milk protein allergy. Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the dry powder inhaler (DPI) (i.e., lactose or magnesium stearate). Historical Allergy: History of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* 12-Lead ECG abnormality: Significant abnormality in the 12-lead electrocardiogram (ECG) performed at screening.
* Tobacco Use: Current smokers or a smoking history of >=10 pack years. A subject may not have used any inhaled tobacco products in the 12 month period preceding the screening visit.
* Previous Participation: Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2014-08-08 (Actual); Study Completion 2014-08-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FEV1 at 15, 30 minutes, 1, 2, 4, 12, 24, 36, 48, 60 and 72 hours post dose. | Baseline (pre dose) and 15, 30 minutes, 1, 2, 4, 12, 24, 36, 48, 60 and 72 hours post dose in each treatment period
  Change from baseline in FEV1 at 15, 30 minutes, 1, 2, 4, 12, 24, 36, 48, 60 and 72 hours post dose. Day 1 Baseline will be defined as Day 1 pre dose measurement for FEV1 for each treatment period.

SECONDARY OUTCOMES:
Time to onset of bronchodilator effect of FF/VI 100/25 mcg | Baseline, 15, 30 minutes, 1, 2, 4 hours post dose in each treatment period
  The time to onset of bronchodilator effect is defined as the time point when FEV1 first meets or exceeds 12% and 200 mL over baseline during the 0-4 hour serial measurements

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116592 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116592?search=study&search_terms=116592#rs
- Available data/document: Clinical Study Report: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register